CLINICAL TRIAL: NCT05503485
Title: Existential Group Treatment for Older Adults (75+) With Psychological Distress in Primary Care: A Randomized Control Trial
Brief Title: Existential Group Treatment for Older Adults (75+) With Psychological Distress in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government); Karlstad University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-06466
Record Dates: First submitted 2022-07-02; First posted 2022-08-16 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Psychological Distress
Keywords: Existential therapy; Existential group therapy; Existential group treatment; Aging; Old adults; Randomized control trial; Anxiety; Depression; Psychological Distress; Primary care
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator
Masking Description: A psychology student will monitor participants self-reported scores for safety reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Existential group treatment (Experimental): Participants who are randomized to the experimental condition will participate in an existential group treatment together with 3 to 6 other participants in seven group sessions of 90-120 minutes each for seven weeks.
  Interventions: Behavioral: Existential group treatment
- Supportive telephone calls (Active Comparator): Participants who are randomized to the control condition will receive brief supportive telephone calls once a week for 7 weeks.
  Interventions: Behavioral: Supportive telephone calls

INTERVENTIONS:
Behavioral: Existential group treatment — The existential group treatment follows a manualised structure focusing on aging-related challenges related to existential themes such as story of life, freedom, loneliness, and death. In order to support patients in finding new, productive ways of engaging in the existential process of aging literary texts, therapy practices and assignments between the sessions are used and each group will be accompanied by two therapists who facilitate the group climate, gently bring the group back on topic and help group members to see different ways of dealing with existential concerns related to aging.
  Other Names: Slottsskogen Existential Group Treatment
  Arms: Existential group treatment
Behavioral: Supportive telephone calls — The supportive caller will provide empathetic basic support, equivalent to the telephone support provided within the Swedish non-governmental organization Mind's "Äldrelinjen". No psychotherapeutic techniques will be applied and there will be no interventions beyond the phone call itself.
  Arms: Supportive telephone calls

SUMMARY:
Symptoms of depression and anxiety are common in older adults, and high suicide rates are observed in this age group in Sweden, as in many countries around the globe. Ageing is accompanied by an increased risk of pain, grief, loss, loneliness, cognitive decline and reduced functional ability, all of which may impact on mental health. Despite these facts, older adults are less likely than their younger counterparts to receive care for their mental health problems.

Within primary care, many older adults with symptoms of depression and anxiety do not fully meet diagnostic criteria for clinical diagnosis. However, these subthreshold states, often conceptualized as "psychological distress" are associated with emotional suffering, reduced quality of life and compromised function in daily life. Psychological distress, which is mainly treated in primary care, has been shown to increase after the age of 65, and to peak at ages 80-89. This points to a need for effective interventions for older adults in primary care to reduce the risk of developing clinical depression and anxiety disorders.

The overall aim of this clinical study is to evaluate, using a randomized control trial design (RCT), an existential psychological group treatment for older adults (75+) with psychological distress in a primary care setting. Research persons randomized to the control arm will receive supportive telephone calls.

Specific research aims include:

1. Do older adults show a) decreased psychological distress, b) decreased experiential avoidance, as well as c) improved quality of life after taking part in existential psychological group treatment? Do those randomized to group treatment have significantly better outcomes compared to those randomized to weekly supportive telephone calls? If so, are the positive effects maintained over time?
2. Is experiential avoidance a mediator in the (potential) reduction of psychological distress?
3. Are there any side effects of existential group treatment/supportive telephone calls?
4. Is an existential psychological group treatment for older adults feasible, based on its fidelity?
5. What are older adults' experiences of participating in the existential psychological group treatment/weekly supportive telephone calls?

DETAILED DESCRIPTION:
In Sweden, psychotherapy is recommended for adults with mild to moderate severity of depression and anxiety. However, studies that target the effectiveness of psychotherapies in older adults are insufficient and seldom conducted according to protocols that take gerontological evidence into account, rendering them less age-appropriate.

The investigators in this research group, recently carried out a focus group study with older adults who had pharmacological treatment for depression. A clear message was that the participants wished for a dialog with their professional caregivers about existential issues. They wanted to talk about thoughts about aging and death. Participants saw death not only as a threat, but also as a potential source of escape from mental pain. The latter echoes our results from our mixed methods study on older adults' reasons for attempting suicide, highlighting the need for older patients with mental health issues to have opportunities for a deeper dialogue with professional caregivers about the existential concerns they experience in daily life as they age.

Existential problems of life such as loneliness and coping with the approach of death and parting have been proposed as central challenges in old age. Interest in these issues is growing, and further catalyzed by the covid-19-pandemic. Existential concerns such as death anxiety and loneliness have been linked to a wide variety of mental health problems and existential therapy is now considered a potential candidate for addressing these problems in a systematic manner. Existential therapy is an established therapy form with roots in the humanistic school of psychology that developed during the 1960's. The therapy aims at helping clients to address and handle existential issues such as meaning, loneliness and death anxiety. Four main schools of existential therapies have been identified, all sharing the main assumption that human life is characterized by inevitable limitations and challenges, and that avoidance and denial of these existential concerns may hinder personal development and contribute to psychopathology. Central themes of human existence commonly addressed in existential therapies including meaning, fear of death and loneliness have recently been linked to subjective wellbeing and psychopathology contributing to a growing interest in existential therapy from therapists practicing other therapy forms such as cognitive-behavioral therapy. Attempts have been made to understand existential concerns in a cognitive-behavioral context.

A meta-analysis on the effect of existential therapy in various patient populations, as well as a quantitative report from primary care both show promising results. However, while existential therapy could be of particular relevance for problems related to aging, the investigators in this research group are aware of no published study in which existential therapy has been adapted specifically for older adult patients with psychological distress. Primary care would be the appropriate setting for such an endeavor.

Design. This is a randomized controlled study in which participants are randomly assigned to a psychological group treatment (7 weeks), or to the control condition (a brief supportive check-in once a week during 7 weeks with a psychology student trained in telephone support). Participants will be block randomized by an independent statistician. The proposed study will follow the CONSORT guidelines. Participants who are randomly assigned to the telephone control group will complete the same evaluations as those participating in the intervention, and at the same points. This design enables us to exclude several alternative explanations, such as time and history, and thus increasing the internal validity of the trial, i.e., the certainty that (potential) effects are the result of the existential group intervention. Since there is little evidence regarding existential group interventions for older adults, using this kind of control group is a first step. A minimum requirement for analyzing mediation (the potential role of experiential avoidance) is a midway measurement.

Therapist training will include study of the treatment manual and simulated training sessions. The following should ensure good implementation of the intervention: 1) treatment manuals with checklists and 2) audio recordings of the group sessions and an evaluation of 25% of these recordings (randomly selected) by an independent evaluator to study the construct validity of the intervention, i.e., whether participants really receive all components included in the intervention.

Recruitment. Older adults (age ≥ 75) with perceived psychological distress residing in the Västra Götalandsregionen are recruited via participating primary care centers.

Screening. Prospective participants will undergo a brief screening comprising a self-report questionnaire on perceived psychological distress, the General Health Questionnaire 12 (GHQ-12). Those with increased levels of psychological distress (GHQ-12 ≥3) will take part in a diagnostic interview with a mental health professional, the Mini-International Neuropsychiatric Interview (M.I.N.I., Diagnostic and Statistical Manual 5 version) and complete a measurement of global cognitive performance (MMSE). The screening can take place at the patient's primary care center or in the home if that is the wish of the potential participant.

Statistical analyses. The investigators will use an intention-to-treat analysis. The data will be analyzed using growth curve models (either with mixed or structural equation modelling) with the aim of examining individual differences and change in variables during and after treatment as well as during the follow-up.Two types of effect measures are of interest. One is the group by time interaction (ie from the pre-intervention measurement to the final measurement, and potentially also the trend deviation between the last session and the 3-month follow-up). The second effect measure is the post-treatment differences between study arms at a) the last session and b) the 3-month follow-up. In combination these should provide a comprehensive evaluation of the (potential) effect of the existential group treatment. If the group treatment has any effect, the investigators will want to examine whether this effect is "driven" by the intervention (interaction effect). The statistical approach is based on regression analyses. Contrary to more traditional variable-oriented analyses for repeated measurements, it has the benefit of better handling missing data, and unbalanced study design, by incorporating all available information. This last method is now regarded as preferable to using more traditional methods for missing data in clinical data. The potential mediator (experiential avoidance) will be examined through different types of regression analyses. To investigate a process such as mediation, at least three points of measurement are needed, and to control for the initial levels of the examined variables.

Power. The investigators in this research group have calculated the number of participants needed, based on earlier studies. Some of these studies showed large effects. However, they involve individual rather than group treatment, and they did not specifically involve older adults, making the results of the meta-analysis less applicable to the current study. Therefore, the investigators choose to calculate power based on a medium effect size. Hence, given a desired power of 0.80 (a 4/5 chance of discovering an effect if it exists, regarded as adequate in this context), a risk level of 5% as well as an effect size of 0.50, 128 participants are needed. Based on participation in the clinical improvement project at Slottsskogen Primary Care Center during 2018-19, the investigators expect a dropout rate of 10%, and thus add another 12 participants (total N=140).

Qualitative analyses of focus group data. The investigators will use focus group interviews to examine older adults' experience of participating in the intervention, with separate focus groups for those with group treatment/telephone support. Focus groups are mainly based on the dynamics that arise in the conversation between group members, which means that the interviewer initiates the topic of the conversation but has a less active role than in individual interviews. There will also be a monitor at each interview to ensure that study topics are covered in accordance with the focus group guide and that all get a chance to participate. The investigators anticipate 8 groups (4 groups per study arm) with a purposive sample of 4-5 participants/group. The focus group interviews will be audio recorded and professionally transcribed. Transcriptions will be analyzed using thematic analysis according to Braun and Clarke. Thematic analysis is about exploring the data material with a focus on recurring meanings, which then form themes.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 75+
2. Have increased levels of psychological distress (GHQ-12 ≥3)
3. Be interested in participating in a research project in which they will receive either group treatment or supportive telephone calls.

Exclusion Criteria:

1. Other ongoing psychological treatment
2. Indications that the group format will be unsuitable due to conditions such as clinical diagnosis of dementia or MMSE ≤25, ongoing severe alcohol use disorder, ongoing post- traumatic stress disorder, ongoing psychotic or manic episodes, or other mental health problems necessitating the offering of other specified treatment, as identified by the M.I.N.I.
3. Inadequate knowledge of Swedish
4. Acute suicide risk according to the M.I.N.I.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Psychological Distress | Pre-intervention, during the intervention (after week 4), immediately after the intervention as well as at a 3-month follow-up
  Measured by General Health Questionnaire (GHQ-12)
Change in Experiential avoidance | Pre-intervention, during the intervention (after week 4), immediately after the intervention as well as at a 3-month follow-up
  Measured by the Brief Experiential Avoidance Questionnaire (BEAQ)

SECONDARY OUTCOMES:
Anxiety symptoms | Pre-intervention, during the intervention (after week 4), immediately after the intervention as well as at a 3-month follow-up
  Measured by the Hospital Anxiety and Depression Scale (HADS)
Depressive symptoms | Pre-intervention, during the intervention (after week 4), immediately after the intervention as well as at a 3-month follow-up
  Measured by the Hospital Anxiety and Depression Scale (HADS)
Zest for life | Pre-intervention, during the intervention (after week 4), immediately after the intervention as well as at a 3-month follow-up
  Measured by the Montgomery-Åsberg Depression Rating Scale-Self report item 9 (MADRS)
Sleep problems | Pre-intervention, during the intervention (after week 4), immediately after the intervention as well as at a 3-month follow-up
  Measured by the Insomnia Severity Index (ISI)
Life quality | Pre-intervention, during the intervention (after week 4), immediately after the intervention as well as at a 3-month follow-up
  Measured by the Brief Quality of Life Scale (BBQ)

OTHER OUTCOMES:
Working Alliance | During the intervention (after week 1 and 4) and immediately after the intervention.
  Measured by the Working Alliance Inventory Short Revised (WAI-SR)
Expectations and credibility of the treatment | During the intervention (after week 1).
  Measured by the Credibility and Expectancy Questionnaire (CEQ)
Side effects | Immediately after the intervention (week 7).
  Measured by the Negative Effects Questionnaire (NEQ)
Group climate | Immediately after the intervention (week 7).
  Measured by questions added to WAI-SR from Robak, R.W., et al. (2013) for participants in the experimental condition.

CONTACTS AND LOCATIONS:
Overall Officials: Margda Waern, Professor, Principal Investigator — Göteborg University
Locations (7):
- Sweden (7):
  - Närhälsan Slottsskogen vårdcentral, Gothenburg
  - Närhälsan Majorna Vårdcentral, Gothenburg
  - Närhälsan Högsbo vårdcentral, Gothenburg
  - Vårdcentralen Wästerläkarna, Gothenburg
  - Capio vårdcentral Orust, Henån
  - Närhälsan Vårgårda vårdcentral, Vårgårda
  - Vårdcentralen Kusten Ytterby, Ytterby

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folkhälsomyndigheten., Skillnader i psykisk ohälsa bland äldre personer: En genomgång av vtenskaplig litteratur samt en epidemiologisk studie. FHM. Stockholm. 2019.
- [Background] Drapeau A, M.A., Beaulieu-Prévost, Epidemiology of psychological distress, in Mental illnesses - understanding, prediction and control. Edited by P. L. Labate, London, Intech Open, pp. 105-34. 2012.
- [Background] Arvidsdotter T, Marklund B, Kylen S, Taft C, Ekman I. Understanding persons with psychological distress in primary health care. Scand J Caring Sci. 2016 Dec;30(4):687-694. doi: 10.1111/scs.12289. Epub 2015 Oct 13. PMID 26463897
- [Background] Cairney J, Krause N. The social distribution of psychological distress and depression in older adults. J Aging Health. 2005 Dec;17(6):807-35. doi: 10.1177/0898264305280985. PMID 16377773
- [Background] Schieman S, Van Gundy K, Taylor J. Status, role, and resource explanations for age patterns in psychological distress. J Health Soc Behav. 2001 Mar;42(1):80-96. PMID 11357720
- [Background] Korte J, Bohlmeijer ET, Smit F. Prevention of depression and anxiety in later life: design of a randomized controlled trial for the clinical and economic evaluation of a life-review intervention. BMC Public Health. 2009 Jul 20;9:250. doi: 10.1186/1471-2458-9-250. PMID 19619284
- [Background] SBU, Statens beredning för medicinsk utvärdering: Behandling av depression hos äldre. En systematisk litteraturöversikt. Stockholm: SBUrapport, 2015, nr: 233.
- [Background] Kishita N, Laidlaw K. Cognitive behaviour therapy for generalized anxiety disorder: Is CBT equally efficacious in adults of working age and older adults? Clin Psychol Rev. 2017 Mar;52:124-136. doi: 10.1016/j.cpr.2017.01.003. Epub 2017 Jan 16. PMID 28119196
- [Background] Rydberg Sterner T, Dahlin-Ivanoff S, Gudmundsson P, Wiktorsson S, Hed S, Falk H, Skoog I, Waern M. 'I wanted to talk about it, but I couldn't', an H70 focus group study about experiencing depression in early late life. BMC Geriatr. 2020 Dec 7;20(1):528. doi: 10.1186/s12877-020-01908-x. PMID 33287708
- [Background] Van Orden KA, Wiktorsson S, Duberstein P, Berg AI, Fassberg MM, Waern M. Reasons for attempted suicide in later life. Am J Geriatr Psychiatry. 2015 May;23(5):536-44. doi: 10.1016/j.jagp.2014.07.003. Epub 2014 Jul 23. PMID 25158916
- [Background] Langle, A. and C. Probst, Existential questions of the elderly. Arch Psychiatry Psychother, 2004. 6(3): p. 15-20.
- [Background] Spitzenstatter D, Schnell T. The existential dimension of the pandemic: Death attitudes, personal worldview, and coronavirus anxiety. Death Stud. 2022;46(5):1031-1041. doi: 10.1080/07481187.2020.1848944. Epub 2020 Dec 24. PMID 33357041
- [Background] Aisenberg-Shafran D, Bar-Tur L, Levi-Belz Y. Who is really at risk? The contribution of death anxiety in suicide risk and loneliness among older adults during the COVID-19 pandemic. Death Stud. 2022;46(10):2517-2522. doi: 10.1080/07481187.2021.1947416. Epub 2021 Jul 19. PMID 34280075
- [Background] Iverach L, Menzies RG, Menzies RE. Death anxiety and its role in psychopathology: reviewing the status of a transdiagnostic construct. Clin Psychol Rev. 2014 Nov;34(7):580-93. doi: 10.1016/j.cpr.2014.09.002. Epub 2014 Sep 22. PMID 25306232
- [Background] Heinrich LM, Gullone E. The clinical significance of loneliness: a literature review. Clin Psychol Rev. 2006 Oct;26(6):695-718. doi: 10.1016/j.cpr.2006.04.002. Epub 2006 Jun 19. PMID 16952717
- [Background] Vos J, Craig M, Cooper M. Existential therapies: a meta-analysis of their effects on psychological outcomes. J Consult Clin Psychol. 2015 Feb;83(1):115-28. doi: 10.1037/a0037167. Epub 2014 Jul 21. PMID 25045907
- [Background] Yalom, I., Existential Psychotherapy. Edited by Basic Books, Library of Congress Cataloging in Publication Data, New York, 1980.
- [Background] Li, J.-B., K. Dou, and Y. Liang, The relationship between presence of meaning, search for meaning, and subjective well-being: A three-level meta-analysis based on the meaning in life questionnaire. J Happ Stud, 2021. 22(1): p. 467-489.
- [Background] Heidenreich T, Noyon A, Worrell M, Menzies R. Existential Approaches and Cognitive Behavior Therapy: Challenges and Potential. Int J Cogn Ther. 2021;14(1):209-234. doi: 10.1007/s41811-020-00096-1. Epub 2021 Jan 4. PMID 33425123
- [Background] Rayner, M. and D. Vitali, Short-term existential psychotherapy in primary care: A quantitative report. J Hum Psychol, 2016. 56(4): p. 357-372.
- [Background] Suri, R., Working with the elderly: An existential-humanistic approach. J Hum Psychol, 2010. 50(2): p. 175-186.
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Folstein MF, Robins LN, Helzer JE. The Mini-Mental State Examination. Arch Gen Psychiatry. 1983 Jul;40(7):812. doi: 10.1001/archpsyc.1983.01790060110016. No abstract available. PMID 6860082
- [Background] Kazdin, A., Methodological issues and strategies in clinical research (fourth edition). American Psychological Association (APA) 2016.
- [Background] Braun, V. and V. Clarke, Using thematic analysis in psychology. Qual res psychol, 2006. 3(2): p. 77-101.